CLINICAL TRIAL: NCT04061005
Title: 7th Medical Center of PLA General Hospital
Brief Title: A Comparison of the Resection Rate for Cold and Hot Snare Polypectomy for 5-15 mm Colorectal Polyps
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yuqi He (Other)
Responsible Party: Sponsor-Investigator, Yuqi He, Principal Investigator, Clinical Professor, General Hospital of Beijing PLA Military Region
Organization: General Hospital of Beijing PLA Military Region (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLA HSP-CSP-1
Record Dates: First submitted 2019-07-29; First posted 2019-08-19 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-02

CONDITIONS: Adenomatous Polyps
Keywords: Cold snare polypectomy; Hot snare polypectomy; Colorectal polyps; CARE Study; Complete resection rate
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Masking Description: RCT-HSP-CSP
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hot snare polypectomy (HSP) (Active Comparator): The polyp size was measured using the tip of the snare catheter (2.5 mm). According to the randomized group, patients with HSP group were treated with HSP to excise 5-15 mm colorectal polyps. After resection, the jet stream will be used to thoroughly clean the mucosal defect. After the endoscopist carefully observed the edge of the resection to complete the polypectomy, a 2- or 4-quad biopsy was performed from the symmetrical margin of the mucosal defect to confirm the presence or absence of residual lesions.
  Interventions: Procedure: Hot snare polypectomy; Procedure: Endoscopic margin observation method
- Cold snare polypectomy (CSP) (Experimental): The polyp size was measured using the tip of the snare catheter (2.5 mm). After randomization, patients in the CSP group will be treated with CSP to remove colorectal polyps of 10-15 mm size. After resection, the jet stream will be used to thoroughly clean the mucosal defect. After the endoscopic surgeon carefully observed the resection margin to complete the polypectomy, a 2- or 4-quad biopsy was performed from the symmetrical margin of the mucosal defect to confirm the presence or absence of residual lesions.
  Interventions: Procedure: Cold snare polypectomy; Procedure: Endoscopic margin observation method

INTERVENTIONS:
Procedure: Cold snare polypectomy — CSP, which does not include electrocautery to do a polypectomy with a snare.
  Arms: Cold snare polypectomy (CSP)
Procedure: Hot snare polypectomy — HSP, which uses the electrocautery to do a polypectomy with a snare.
  Arms: Hot snare polypectomy (HSP)
Procedure: Endoscopic margin observation method — Endoscopic margin observation method, After rinsing the polyp specimen with physiological saline, fully natural extension, fixing it to the foam board with a needle, and observing the margin with a colonoscope or a magnifying colonoscope near-focus mode to determine whether there is residual polyp tissue.

SUMMARY:
In 2015, there were approximately 1.7 million new cases of colorectal cancer（CRC）, and the deaths was close to 832,000. CRC has become the third most common malignant tumor in the world and the second leading cause of cancer death. This is mainly because adenomatous polyps can be transformed into cancer through adenoma-cancer sequences. Screening for CRC has been shown to prevent CRC and related deaths, especially colonoscopy and endoscopic resection of adenomatous polyps.

Currently, the main methods of resection for polyps below 20 mm include hot snare polypectomy (HSP) and cold snare polypectomy (CSP). Due to the use of electrocautery, HSP has been shown to cause damage to the deep submucosa, the muscularis propria and submucosal arteries, resulting in postoperative bleeding, perforation and other adverse events. Compared with HSP, the mechanical cutting method is called CSP without electrocautery. Due to the short operation time and low incidence of adverse events, especially after polypectomy, it has caused more and more attention of endoscopists. The removal of 5 mm polyps from CSP has been recommended as the preferred technique by the European Society of Gastrointestinal Endoscopy(ESGE) Guidelines. A recent multicenter, prospective study in Japan recommended CSP as the standard treatment for excision of 4-9mm polyps. However, the average diameter of polyps in this study was 5.4 mm, which was not sufficient for the safety of CSP in polyps above 5 mm. In addition, there are few prospective studies of CSP complete removal of colorectal polyps 10-15 mm. More importantly, the report pointed out that 10% of 5 to 20 mm polyps were not completely removed, and some studies have shown that the cut polyp specimens are not sufficient for adequate pathological evaluation, which the researchers do not fully recognize.

In this study, the investigators were interested in comparing the complete resection rates of large (10 -15 mm) and small (4-9 mm) colorectal polyps with CSP and HSP and improved methods for evaluating complete resection.

DETAILED DESCRIPTION:
Participants who meet inclusion criteria will be asked to participate, investigators will include all patients with resectable polyps, but only adenomatous polyps will be included for analysis. See also inclusion and exclusion criteria.

Colonoscopy, after bowel preparation with polyethylene glycol solution was performed using standard colonoscopes (GIF-HQ290I) and polypectomy snares.

All procedures were performed by experienced endoscopists(each with over 1000 colonoscopies performed) including CSP and HSP. All patients with a colorectal 5-15 mm polyp detected will be randomized to receive HSP and CSP treatment. Polyp size will be measured using the tip of the snare catheter (2.5mm). Difficulty of resection will be grade by polyp resection time. Following the resection, jet stream of water will be used to wash mucosal defect thoroughly. After endoscopist's attestation that polyp removal was complete by carefully observe the resection margins with near focus mode, for large lesions(10-15mm)4 biopsies will be performed from all four quadrants of resection margins, for small lesions(4-9mm) biopsies were performed from two marginal sites located symmetrically on the left and right of the mucosal defects to confirm residual polyp tissue. Difficulty of resection will be grade by polyp resection time. Following the resection, jet stream of water will be used to wash mucosal defect thoroughly. After endoscopist's attestation that polyp removal was complete by carefully observe the resection margins with near focus mode, for large lesions(10-15mm)4 biopsies will be performed from all four quadrants of resection margins, for small lesions(4-9mm) biopsies were performed from two marginal sites located symmetrically on the left and right of the mucosal defects to confirm residual polyp tissue.

If polyp resection is complicated by bleeding(not self-sustained), no biopsies will be taken and any additional polyps that will be found during the remaining examination will be excluded from analysis. Severe bleeding that will complicate resection margins examination will be excluded from analysis, Endoscopic haemostasis will be performed when active haemorrhage continued for ≥30s.

A single research subject may have many eligible polyps. To avoid taking many biopsies, the investigators will not include more than 5 eligible polyps(the first 5 that are detected) per patient in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥40 and <70 years old
* Provide written informed consent
* Patients are found to have colorectal polyps between 5 and 15mm in size

Exclusion Criteria:

* History of inflammatory bowel disease
* Polyposis of the alimentary tract
* Antiplatelet or anticoagulant therapy 5 days before the procedure
* Pregnancy
* Haemodialysis
* An American Society of Anaesthesiologists class III or higher
* Depressed lesions and lesions highly suspected to be cancerous based on endoscopic appearance.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2018-08-20 (Actual); Primary Completion 2022-10-20 (Estimated); Study Completion 2022-10-20 (Estimated)

PRIMARY OUTCOMES:
Complete resection rate | six months
  The primary endpoint was the complete resection rate, defined as no evidence of adenomatous tissue in the biopsied specimens, among all pathologically confirmed adenomatous polyps. The complete resection rates in the HSP and CSP groups of 5-15mm polyps were compared. The complete resection rates in the HSP and CSP groups of 5-9 mm polyps group were compared. and the complete resection rates in the HSP and CSP groups of 10-15 mm polyps group were also compared.

SECONDARY OUTCOMES:
Methodological evaluation of Endoscopic margin observation method | six months
  After polypectomy, the operating assistant unfolded the retrieved polyp specimen in the natural shape and pinned flat on a cork board according to the ESD specimen fixation method. Then endoscopic view judged the margin of the unfolded polyp.If a complete normal mucosal margin is visible, it is considered a complete resection. Then, the complete resection rate of the method was compared with the complete resection rate of the traditional pathological biopsy to judge the accuracy of the method.
Polyp retrieval rate | six months
  Polyp specimens retrieval rate
Number of additional resections (snaring and/or biopsy) | six months
  snaring and/or biopsy
Rate of difficult/impossible resection by CSP | six months
  Difficult CSP resection was defined as a resection procedure that required ≥5s after snaring.An impossible CSP resection was defined as a resection procedure that needed high-frequency electric current.
Time required for resection | six months
  Time required for resection was defined as the time between the insertion of the snare into working channel to the end of polyp resection. The time was measured by endoscopists or assistant by using stopwatch that was built in the endoscopic system. When submucosal injection was conducted in the HSP group, the time required for resection was measured from the insertion of the injection needle into the working channel until the end of polyp resection.
The rates of procedure-related complications | six months
  Delayed bleeding was defined as haemorrhage after colonoscopy requiring endoscopic haemostasis. It should be noted that, if vascular stump is found on the wound surface after HSP, electrocoagulation treatment is required and the probability is recorded.After CSP, it is necessary to observe whether there is active bleeding.Titanium clips were not used for hemostasis in both groups.

CONTACTS AND LOCATIONS:
Overall Officials: tianyang zhang, Principal Investigator — Medical department
Locations (1):
- Department of Gastroenterology, 7th medical center of PLA general hospital, Beijing, Dongcheng District, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kawamura T, Takeuchi Y, Asai S, Yokota I, Akamine E, Kato M, Akamatsu T, Tada K, Komeda Y, Iwatate M, Kawakami K, Nishikawa M, Watanabe D, Yamauchi A, Fukata N, Shimatani M, Ooi M, Fujita K, Sano Y, Kashida H, Hirose S, Iwagami H, Uedo N, Teramukai S, Tanaka K. A comparison of the resection rate for cold and hot snare polypectomy for 4-9 mm colorectal polyps: a multicentre randomised controlled trial (CRESCENT study). Gut. 2018 Nov;67(11):1950-1957. doi: 10.1136/gutjnl-2017-314215. Epub 2017 Sep 28. PMID 28970290
- [Result] Matsuura N, Takeuchi Y, Yamashina T, Ito T, Aoi K, Nagai K, Kanesaka T, Matsui F, Fujii M, Akasaka T, Hanaoka N, Higashino K, Tomita Y, Ito Y, Ishihara R, Iishi H, Uedo N. Incomplete resection rate of cold snare polypectomy: a prospective single-arm observational study. Endoscopy. 2017 Mar;49(3):251-257. doi: 10.1055/s-0043-100215. Epub 2017 Feb 13. PMID 28192823